CLINICAL TRIAL: NCT06197048
Title: A Randomized Controlled Trial on the Effect of Nutritional Counseling on Anthropometry and Biomarkers in Patients Diagnosed With Schizophrenia/Psychosis or Bipolar Affective Disorder Treated at Asker DPS as Outpatients or Inpatients at Blakstad Hospital
Brief Title: Effect of Nutritional Counseling on Anthropometry and Biomarkers in Patients Diagnosed With Schizophrenia/Psychosis or Bipolar Affective Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Vestre viken
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Diseases; Schizophrenia; Psychosis; Bipolar Disorder
Keywords: Severe mental disorders; Nutritional counseling; Cardiovascular disease; Schizophrenia; Bipolar affective disorder; Randomzied controlled trial
MeSH Terms: conditions — Cardiovascular Diseases; Schizophrenia; Psychotic Disorders; Bipolar Disorder; Mental Disorders | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: the included patients will be randomized into two groups: one croup will receive nutritional counseling, while the other does not. All the participants will complete baseline and post-intervention measurements consisting of: mapping of diet, anthropometric measurements (weight, height, waist measurement), bloodpressure, biochemical measurements (total cholesterol, non-HDL cholesterol, LDL cholesterol, triglycerides, vitamin D, ferritin, fasting glucose, HbA1c, folate and AST/ALT. Then the two groups will be compared to reveal any differences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Nutritional counseling — The intervention group will recieve 30 x 2 minutes with nutritonal counseling seperatet by a 15 minutes break. The participants will receive individually tailored guidance based on the information recieved at baseline measurments.
  The couseling will be based on the Norwegian goverments dietary advices and the recommendation from the Directorate of Health for the prevention of cardiovascular diseases.

SUMMARY:
The goal of this clinical trial is to compare the effect of nutritional counseling versus no treatment in patients with schizophenia or bipolar affective disorder.

The main question it aims to answer are:

• Can nutritional counseling have a preventive effect on the development of cardiovascular disease in patients with schizophenia or bipolar affective disorder?

Participants will meet a nutritionist at baseline to asess nutritional status, biochemical and anthropometric measurements. Then, half of the study population will receive nutritional counseling. After six weeks, the same baseline measurements will be repeated to examine any potential differences between the two groups. After the intervention, the control group will be offered the same counseling as the intervention group received during the study.

DETAILED DESCRIPTION:
People with severe mental illness have a shorter life expectancy compared to the general population. Individuals with schizophrenia or bipolar affective disorder have an estimated reduce life expectancy by an average of 10-20 years. Increased mortality is caused by many factors, but cardiovascular diseases contributes the most. Increased prevalence of cardiovascular disease is mainly due to a poor lifestyle, which includes smoking, physical inactivity and an unhealthy diet.

It is important to find treatment that can provide better quality of life and longer life expectancy in these patient groups. Few clinical studies have been conducted on the effect of nutritional counseling on biochemical and anthropometric measurements related to cardiovascular diseases. Therefore, we want to investigate this through a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Diagnosed with either schizophrenia/psychosis or bipolar affective disorder
* Patients treatet in Vestre Viken healthcare company, at either Asker district psychiatric center or Blakstad hospital

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Non-HDL cholesterol | 6 weeks
  HDL-cholesterol - total cholesterol, biochemical test

SECONDARY OUTCOMES:
total cholesterol | 6 weeks
  biochemical test
HDL-cholesterol | 6 weeks
  biochemical test
Triglycerids | 6 weeks
  biochemical test
HbA1c | 6 weeks
  biochemical test
ALT AST/ALT AST/ALT | 6 weeks
  biochemical test
fasting glucose | 6 weeks
  biochemical test
Vitamin D | 6 weeks
  biochemical test
Folate | 6 weeks
  biochemical test
LDL-cholesterol | 6 weeks
  biochemical test
Weight | 6 weeks
  anthropometric measurement
waist circumference | 6 weeks
  anthropometric measurement
Bloodpressure | 6 weeks
24-hour dietary recall | 6 weeks
  interview
Food frequency questionnaire | 6 weeks
  questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Vestre Viken Health Trust, Drammen, Akershus
  - Department of Research and Delvelopment, Mental health and Addiction, Vestre Viken Hospital Trust, Drammen

IPD SHARING:
Plan to Share IPD: No
The IPD will be stored at TSD- services for sensitive data. Only researchers in this prosject will have acsess